CLINICAL TRIAL: NCT03938870
Title: CNS Tau Kinetics in Healthy Aging and Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: BrightFocus Foundation (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 201502091
Record Dates: First submitted 2015-06-22; First posted 2019-05-06 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer's Disease; Brain Diseases; Central Nervous System Diseases; Delirium, Dementia, Amnestic, Cognitive Disorders; Dementia; Mental Disorders; Nervous System Diseases; Neurodegenerative Diseases; Tauopathies
Keywords: Alzheimer's Disease; Alzheimer's; biomarker; dementia; Tau; Tau Kinetics; Tauopathies
MeSH Terms: conditions — Alzheimer Disease; Brain Diseases; Central Nervous System Diseases; Neurocognitive Disorders; Dementia; Mental Disorders; Nervous System Diseases; Neurodegenerative Diseases; Tauopathies; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and Cerebrospinal Fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Experimental: Group 1: 30 Young Normal Controls(YNC) ages 18 & Older will enroll to evaluate leucine infusion methods of labeling, vs. the oral method. They will have 5 lumbar punctures (LPs) and the amount of labeled tau in the CSF will be analyzed to obtain tau kinetics in human central nervous system (CNS).
  Interventions: Other: L-Leucine 13C6
- Experimental: Group 2: Group 30 CDR > 0. There will be collection of CSF and blood. The participants will either be labeled by intravenous infusion method with leucine or oral method based off the results from the Young Normal Control Group. They will have 5 lumbar punctures (LPs) and the amount of labeled tau in the CSF will be analyzed to obtain tau kinetics in human central nervous system (CNS).
  Interventions: Other: L-Leucine 13C6
- Experimental: Group 3: Group of 40 CDR = 0 Age Matched. There will be collection of CSF and blood. The participants will either be labeled by intravenous infusion method with leucine or oral method based off the results from the Young Normal Control Group. They will have 5 lumbar punctures (LPs) and the amount of labeled tau in the CSF will be analyzed to obtain tau kinetics in human central nervous system (CNS).
  Interventions: Other: L-Leucine 13C6

INTERVENTIONS:
Other: L-Leucine 13C6

SUMMARY:
Alzheimer's disease (AD) is the most common cause of dementia and currently has no disease modifying treatments or simple accurate diagnostic tests. The goal of this project is to study how tau (a protein thought to cause AD) is made, transported and cleared in the human body. Better understanding of these processes may lead to improved understanding of AD, earlier diagnosis and a way to evaluate treatment.

DETAILED DESCRIPTION:
The goal of this study is to examine how tau works in the Human Central Nervous System (CNS)and to test the hypothesis, that tau is altered (i.e. increased production, decreased clearance, and increased collection rate) with age, and in diseases caused by the disruption of how tau usually works. We will first test this hypothesis in AD and then test and compare other tau diseases in future studies. We have recently developed a novel approach to measure tau in the human CNS. We propose to utilize this approach to address fundamental questions of human tau production and metabolism in Alzheimer's disease. Researchers have designed this study to determine how long tau stays in the body. It involves labeling or marking tau with a special type of an essential amino acid called leucine. Our bodies naturally get leucine from the foods that we eat.

In this study, the participant will either be given labeled leucine through intravenous infusion, or be given labeled leucine in a drink. The researchers think that it would be more convenient for the participant if the study was done giving the leucine by infusion but this method has not been tested with tau. The first part of the study is to test the infusion method and find the optimal infusion rate and length of time to hopefully see tau. If the method cannot be confirmed with the young normal control group the study will move on to using the oral method of labeling. This has been proven to work but it will be more burdensome for the participants. The leucine is a stable form of carbon found in nature and has no side effects but it will stick to certain proteins such as tau making the tau "visible" to researchers. Once labeled, the researchers will take samples of Cerebral Spinal Fluid (CSF) at different time points and determine how long the tau stays in the system. This amount of time is called the "half-life". Knowing the half-life of tau will help researchers to develop clinical trials that target tau and future therapeutic interventions for AD.

The first type of labeling is Intravenous Infusion of Leucine. After successful screening, the subject would come to the CARS at 07:00 AM, (fasting from 10:00 PM the night before), and have an intravenous catheter placed. The researchers do not know exactly how much Leucine it will take to successfully label Tau so that they can see it. The first studies will be with Young Normal controls ages 18 and older. The researcher will test the following amounts of leucine; Leucine infusion for 24 hours at a rate of 4 mg/kg/hour. The researchers will process the samples immediately. If tau is visible at this amount a second participant will receive a lesser infusion time, leucine infusion for 16 hours at a rate of 4mg/kg/hour. The researchers will process the samples immediately, if tau is visible at this amount a third participant will receive a lesser amount of leucine to label tau. Leucine infusion at a rate of 2/mg/kg/hour for 24 hours. The samples will be tested and if the tau is seen at this amount then a lesser amount of infusion time will be tried. The leucine infusion will be done at at rate of 2/mg/kg/hour for 16 hours. This would be the goal of the study to infuse the least amount of leucine for the least amount of time.

All meals are prepared by the Research Kitchen. When receiving leucine the participant has to have their meals controlled for the natural leucine found in our diets. The participant receives three meals and three snacks in the 24 hours and then a BJC cafeteria breakfast after their first lumbar puncture.

Once the amount and time of leucine infusion is optimal more Young Normal Controls will repeat the infusion study for confirmation. Each participant will complete a total of 5 Lumbar Punctures over time.

If the infusion method is not capable of showing adequate levels of tau the study will move on to the Oral method of labelling. Participants will come to the Research Kitchen on day one to pick up meals for two days, leucine for two days, as well as a diet diary. Participants will receive a great deal of explanation and support as this method is burdensome because of the visits, three days a week to pick up their food, as well as needing to mix, and drink leucine in Kool-Aid 3 times a day for 10 days, and keep a diet diary.

Once participants are labeled the Lumbar Punctures are performed. The Infusion and the Oral method each have a schedule of Lumbar Puncture days.

Fundamental questions of tau kinetics and processing have not been addressed in humans. There has been no reliable technique to measure in vivo tau metabolism. Questions such as 1)what is the half-life of tau in the human central nervous system (CNS), 2)is cerebrospinal fluid (CSF) tau increased due to over-production or under-clearance, 3)are tau kinetics altered in Alzheimer's Disease (AD), and 4)how much should tau be modulated by drugs which target tau have not been addressed to date in humans. We propose to apply a recently developed tau stable isotope labeling kinetics (SILK) method to measure tau kinetics in AD patients and age-matched cognitively normal controls to determine physiological and pathophysiological changes in tau metabolism. We hypothesize that tau production will be increased in AD.

Aim 1: To measure physiological tau kinetics with the tau SILK method in the CNS of normal human participants and determine the effects of age. (a) We will quantify in vivo CNS tau SILK kinetics of 10 YNCs (Age 18-64) and determine the physiological kinetics of human tau. (b) We hypothesize that tau half-life and clearance are slowed with increasing age. Tau kinetics under normal physiological conditions will be compared across different age groups. The participants with normal CSF tau concentrations and normal tau PET imaging results from 10 age-matched controls (age 65 and greater) from Aim 2 will be included in the analyses.

Aim 2: To determine pathological changes in tau kinetics in AD dementia. We hypothesize that soluble tau production is increased in AD with subsequent increase in aggregation rates and irreversible loss of soluble tau. We will examine the kinetics of CNS tau in 10 participants with late-onset AD dementia and 10 cognitively normal age-matched controls (age 65 and greater).

Results from this tau SILK study will help elucidate the dynamic kinetics of human CNS tau in physiology and pathophysiology of tauopathies. The tau SILK method will facilitate future efforts to evaluate the efficacy of tau-targeted therapies and help effectively design future

Genetic and biochemical evidence suggest that amyloid beta and tau contribute to the pathogenesis and pathophysiology of Alzheimer's Disease(AD). Tau cerebral spinal fluid (CSF) levels correlate with cognitive decline in AD, but currently we have little knowledge of tau metabolism in humans as no prior method could test the hypothesis that kinetics of tau are altered in disease. We pioneered the Stable Isotope Labeling Kinetics (SILK) to determine Abeta; kinetics and demonstrated increased Abeta42 production in mutation carriers of early onset AD and decreased Abeta; clearance in sporadic AD. We now propose to use recently developed tau SILK method to determine the tau kinetics in human central nervous system (CNS). Previous studies using mouse models suggest that tau is a slow turnover protein with a half-life of approximately 2 weeks. It is also less abundant compared to Abeta; however, we have utilized sensitive mass spectrometry method to detect and measure labeled tau in human CSF.

Quantitation of the physiological and pathological kinetics of tau in this proposal will be crucial for understanding the pathogenesis of AD and other tauopathies. For example, questions such as 'why is tau increased in AD CSF - overproduction or impaired clearance?' need to be addressed to guide therapeutic targeting. By quantifying the changes in tau production and clearance, better estimates of target engagement can be made. The tau SILK method will be an invaluable tool in future studies to determine the pathophysiology of tau in AD and other neurodegenerative diseases (e.g. Corticobasal degeneration (CBD), Progressive supranuclear palsy (PSP), and Frontotempral Dementia (FTD)) and to evaluate potential drug candidates and genetic manipulations which target Tau. A combination of the tau SILK protocol and a novel tau PET (T807) imaging allows us to examine in-depth the in vivo human soluble and aggregate tau dynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of any race aged 18 or older
2. No evidence of a neurologic disorder or traumatic head injury by history or examination
3. Able to take food and drink by mouth safely
4. Participants must be able to provide informed consent
5. Absence of exclusion criteria

Exclusion Criteria:

1. Requires tube feeding for nutrition and/or hydration
2. Already on a special diet (e.g. Gluten free)
3. History of bleeding disorder
4. Allergy to Lidocaine
5. Pregnancy
6. Any contraindication for lumbar puncture e.g. blood thinners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will recruit 100 participants (age 18+) 30 Young Normal Controls, 30 AD participants (age 65+) and 40 age-matched controls (age 65+) to participate in this study. Studies will be conducted at the Clinical Trials Research Unit at Washington University School of Medicine. Volunteers will be screened for any major medical abnormalities, bleeding risks, or any other reason they might not tolerate the procedure.
  The participants will either be labeled by intravenous infusion method or oral method. They will have 5 lumbar punctures (LPs) and the amount of labeled tau in the CSF will be analyzed to obtain tau kinetics in human central nervous system (CNS).
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Tau kinetics in cerebrospinal fluid [half-life of tau], as assessed by tau stable isotope labeling kinetics (SILK) method | 4 months
  To measure physiological tau kinetics with the tau SILK method in the CNS of human participants.

SECONDARY OUTCOMES:
Age | 4 months
  Physiological tau kinetics in CNS will be analyzed to determine the effects of age.
Tau aggregation measured by PET Imaging | 4 months
  Correlation between tau kinetics (SILK) measures [half-life of tau] and Tau PET Imaging results will be assessed.
Amyloid aggregation measured by PET Imaging | 4 months
  Correlation between tau kinetics (SILK) measures [half-life of tau] and Amyloid PET Imaging results will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Bateman, MD, Principal Investigator — Washington University in Saint Louis
Locations (1):
- Washington University in Saint Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bateman RJ, Munsell LY, Morris JC, Swarm R, Yarasheski KE, Holtzman DM. Human amyloid-beta synthesis and clearance rates as measured in cerebrospinal fluid in vivo. Nat Med. 2006 Jul;12(7):856-61. doi: 10.1038/nm1438. Epub 2006 Jun 25. PMID 16799555